CLINICAL TRIAL: NCT07348328
Title: Vitamin B Supplementation for Patients Undergoing Cardiovascular Surgery: A Randomized Controlled Trial
Brief Title: Vitamin B Supplementation for Patients Undergoing Cardiovascular Surgery
Acronym: PANDA XII
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); West China Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Department of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PANDA XII
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Surgical Procedures; Major Adverse Cardiovascular Events (MACE)
Keywords: Compound Vitamin B; Cardiovascular Surgery; Major Adverse Cardiovascular Events

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B supplementation (Experimental): perioperative supplementation with Compound Vitamin B tablets, once daily from 3 days before surgery to 6 months after surgery
  Interventions: Drug: Compound Vitamin B tablet
- Control (Placebo Comparator): perioperative supplementation with oral placebo, once daily from 3 days before surgery to 6 months after surgery
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Compound Vitamin B tablet — perioperative supplementation with Compound Vitamin B tablets, once daily from 3 days before surgery to 6 months after surgery
  Arms: Vitamin B supplementation
Drug: Control — perioperative supplementation with placebo, once daily from 3 days before surgery to 6 months after surgery
  Arms: Control

SUMMARY:
This study is a multicenter, randomized controlled, double-blind, placebo-controlled parallel trial designed to evaluate the effect of perioperative supplementation with Compound Vitamin B on patients undergoing cardiovascular surgery. A total of 1,000 patients aged 18-80 years who are scheduled to receive cardiovascular surgeries such as coronary artery bypass grafting (CABG) and valve replacement will be enrolled. They will be randomly assigned at a 1:1 ratio to either the experimental group (perioperative supplementation with Compound Vitamin B tablets, once daily from 3 days before surgery to 6 months after surgery) or the control group (oral placebo), with both groups receiving standardized perioperative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years, regardless of gender;
* Scheduled to receive cardiovascular surgery at the research center, including coronary artery bypass grafting (CABG), cardiac valve replacement/repair, and great vessel surgery;
* Preoperative assessment indicates that the patient is expected to complete the 6-month postoperative follow-up;
* The patient or their authorized agent signs a written informed consent form.

Exclusion Criteria:

* Regular supplementation with Compound Vitamin B (daily dose ≥ 1.5 times the recommended dietary allowance) or separate supplementation with folic acid, vitamin B6, or B12 within 3 months before surgery;
* Severe hepatic or renal insufficiency (liver function: ALT/AST > 3 times the upper limit of normal, or total bilirubin > 2 times the upper limit of normal; renal function: serum creatinine > 265 μmol/L, or requiring long-term dialysis treatment);
* Malignant tumors, severe hematological diseases (e.g., megaloblastic anemia, aplastic anemia), severe malnutrition (albumin < 25 g/L);
* History of allergy to Compound Vitamin B preparations or placebo components; Pregnant women, lactating women, or those planning to become pregnant during the study period;
* Currently participating in other interventional clinical trials;
* Moderate to severe cognitive impairment without a fixed caregiver, unable to cooperate with treatment and follow-up;
* Preoperatively diagnosed with severe infection, septicemia, or septic shock.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the incidence of MACE | within 6 months after surgery between the two groups
  MACE is defined as a composite endpoint, including: cardiac death, non-fatal myocardial infarction (postoperative troponin peak > 10 times the upper limit of normal accompanied by chest pain and dynamic changes in electrocardiogram), ischemic stroke (new-onset neurological deficits after surgery confirmed by cranial CT/MRI), severe arrhythmia (sustained ventricular tachycardia, ventricular fibrillation, third-degree atrioventricular block requiring implantation of a temporary/permanent pacemaker), and readmission due to cardiac causes.

CONTACTS AND LOCATIONS:
Overall Officials: Guo-liang Fan, Study Chair — Shanghai East Hospital
Locations (2):
- China (2):
  - Shanghai East Hospital Tongji University, Shanghai, DR
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing

IPD SHARING:
Plan to Share IPD: Undecided